CLINICAL TRIAL: NCT01575561
Title: A Multi-center, Open Label, Flexible Dose, Extension Study of Lurasidone Adjunctive to Lithium or Divalproex in Subjects With Bipolar I Disorder
Brief Title: This is an Open-label, Multi-center, Extension Study Designed to Evaluate the Longer Term Safety, Tolerability and Effectiveness of Lurasidone, Flexibly Dosed, Adjunctive to Lithium or Divalproex for the Treatment of Subjects With Bipolar I Disorder Who Have Participated in Study D1050296
Acronym: PERSISTExt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1050308; 2011-004789-14 (EudraCT Number)
Record Dates: First submitted 2012-03-28; First posted 2012-04-11 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Bipolar I Disorder
Keywords: Lurasidone; Latuda; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lurasidone (Experimental): Lurasidone 20, 40, 60,80 mg flexible dose
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Lurasidone 20-80 mg taken orally once daily

SUMMARY:
This is an open-label, multi-center,12 week extension study designed to evaluate the longer term safety, tolerability and effectiveness of lurasidone, flexibly dosed, adjunctive to lithium or divalproex for the treatment of subjects with bipolar I disorder, who have either completed the core study D1050296 or experienced a protocol defined recurrence of a mood event in the double-blind phase of the core study D1050296

DETAILED DESCRIPTION:
To evaluate the longer term safety of lurasidone (20, 40, 60 or 80 mg/day) in subjects with bipolar I disorder.

Subjects will be initially treated with open-label lurasidone 40 mg/day (Day 1).

Dose adjustment of study drug (20, 40, 60 or 80 mg /day) should occur at the regularly scheduled visits and in increments/decrements of 1 dose level.

ELIGIBILITY:
Inclusion Criteria:

* Subject has agreed to participate by providing written informed consent.
* Subject has completed the 28 week Double-blind Phase of Study D1050296 and all required assessments on the final study visit (Week 28, Visit 28); OR
* Subject has experienced a protocol-defined recurrence of any mood event during the Double blind Phase of Study D1050296 and has completed all required assessments on the final study visit; OR
* Subject had at least entered the Open-label Phase of Study D1050296 when the Sponsor stopped the study and has completed all required assessments on the final study visit.
* Subject is judged by the Investigator to be suitable for participation in a 12 week clinical trial involving open-label lurasidone treatment and is able to comply with the protocol in the opinion of the Investigator.

Exclusion Criteria:

* Subject is considered by the Investigator to be at imminent risk of suicide or injury to self, others, or property.
* Subject answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the Columbia Suicide Severity Rating Scale (C-SSRS) at the extension baseline visit (final study visit in Study D1050296).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2012-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lurasidone Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (70):
- United States (25):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Behavioral Research Specialists, LLC, Glendale, California
  - AXIS Clinical Trials, Los Angeles, California
  - Excell Research, Inc, Oceanside, California
  - Stanford University School of Medicine Research Program VA Palo Alto Health Care System, Palo Alto, California
  - SF-Care, Inc., San Francisco, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Stanford University School of Medicine, Stanford, California
  - Florida Clinical Research LLC, Bradenton, Florida
  - Clinical Neuroscience Solutions Inc., Jacksonville, Florida
  - Galiz Research, Miami Springs, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Clinco, Terre Haute, Indiana
  - Activ Med Practices & Research, Haverhill, Massachusetts
  - Psych Care Consultants Research, St Louis, Missouri
  - Finger Lakes Clinical Research, Rochester, New York
  - Charak Clincial Research Center, Garlield Heights, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Carolina Clinical Trials, Charleston, South Carolina
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Psychoneuroendocrinology Research Group, Dept of Psychiatry, UT Southwestern Medical Center, Dallas, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
- Argentina (6):
  - Clinica Privada de Salud Mental Santa Teresa de Avila, Buenos Aires
  - Novain Neurociencias Group, Buenos Aires
  - Instituto Nacional de Psicopatología (INAPSI), Buenos Aires
  - Fundacion para el estudio y tratamiento de las enfermedades mentales (FETEM), Buenos Aires
  - Instituto DAMIC SRL, Córdoba
  - Centro de Investigacion y Asistencia en Psiquiatria (CIAP), Rosario
- Bulgaria (3):
  - Center for Mental Health, Rousse
  - Multiprofiled Hospital for Active Treatment "Alexandrovska", Sofia
  - Military Medical Academy, Sofia
- Chile (2):
  - Hospital El Pino, Santiago
  - Clinica Pedro Montt, Santiago
- Czechia (7):
  - Saint Anne, s.r.o., Psychiatricke oddeleni, Brno - Mesto
  - Psychiatricka ambulance, Havířov
  - Psychiatricka lecebna U Honzicka, Písek
  - Clintrial s.r.o., Prague
  - Psychiatricka ambulance, Prague
  - Psychiatricka ambulance Prosek, Prague
  - Telemens, s.r.o., Přerov
- France (3):
  - CHS La Chartreuse - Pôle 6, Dijon
  - Centre Hospitalier Spécialisé du Jura - Centre Médico Psychiatrique, Dole
  - Centre Hospitalier Régional Universitaire, Nîmes
- Hungary (4):
  - Kutvolgyi Klinikai Tomb SOTE IIIsz Belgyogyaszati Klinika, Budapest
  - Nyiro Gyula Korhaz, I. Pszichiatria, Budapest
  - Nyiro Gyula Korhaz, II. Pszichiatria, Budapest
  - Nyiro Gyula Korhaz, Budapest
- Japan (5):
  - Goryokai Medical Corporation, Sapporo, Hokkaido
  - Asakayama General Hospital, Sakai, Osaka
  - Yuge Hospital, Kumamoto
  - Nishigahara Hospital, Tokyo
  - Kawada Hospital, Toyama
- Poland (3):
  - NZOZ Syntonia, Gdynia
  - NZOZ BioMed, Kielce
  - NZOZ Prywatna Klinika Psychiatryczna Inventiva, Tuszyn
- Russia (6):
  - State Healthcare and Forensic Psychiatric Expertise Institution, Izhevsk
  - Saint Petersburg State Healthcare Institution "City psycho-neurology Dispanser #7", Saint Petersburg
  - St Petersburg State Government Healthcare Institution, Saint Petersburg
  - St. Petersburg State Healthcare Institution "City Clinical Hospital #4", Saint Petersburg
  - Mental Health Research Institute of Siberian Branch of RAMS, Tomsk
  - Nizhny Novgorod Regional State Institution of Healthcare, Veliky Novgorod
- Serbia (4):
  - Clinical Hospital Centre Dragisa Misovic, Belgrade
  - Clinical Centre Kragujevac, Psychiatric Hospital, Kragujevac
  - Clinic for Mental Health Protection, Clinical Centre Nis, Niš
  - Specialized Hospital for Psychiatric Diseased "Sveti Vracevi", Novi Kneževac
- Slovakia (2):
  - Psychiatricke oddelenie, Vseobecna nemocnica Rimavska Sobota NaP n.o., Rimavská Sobota
  - Psychiatricka ambulancia, Zlaté Moravce

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lurasidone
Started | 377
Completed | 338
Not Completed | 39
Not completed — Adverse Event | 9
Not completed — Lack of Efficacy | 8
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 11
Not completed — administration | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lurasidone
Number analyzed (Participants) | 377
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 359
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62
  Not Hispanic or Latino | 315
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 327
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  Czech Republic | 40
  Russian Federation | 42
  Argentina | 30
  Hungary | 21
  United States | 95
  Japan | 13
  Poland | 37
  Slovakia | 5
  Bulgaria | 34
  France | 8
  Chile | 17
  Serbia | 35

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events and Treatment-emergent Adverse Events Leading to Discontinuation and Serious Adverse Events
Description: Number of subjects with treatment emergent AEs, SAEs, and TEAEs leading to discontinuation
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Lurasidone
Number analyzed (Participants) | 377
participants
  at Least 1 TEAE potentially related to study drug | 155
  subjects with at least one TEAE potentially relate | 69
  at least 1 treatment emergent SAE | 14
  at least 1 treatment emergent SAE related to drug | 1
  at least 1 TEAE leading to discontinuation | 9

2. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the Quick Inventory of Depressive Symptomatology - Self Report (QIDS SR16) Total Score
Description: The QIDS-SR16 is a 16-item self-report measure of depressive symptomatology which uses a computerized assessment interface for administration. The scoring system for the QIDS-SR16 converts responses to 16 separate items into nine DSM-IV symptom criterion domains. The nine domains comprise: depressed mood (Item 5); concentration/decision making (Item 10); self outlook (Item 11); suicidal ideation (Item 12); decreased interest (Item 13); decreased energy (Item 14); sleep disturbance (initial, middle, and late insomnia or hypersomnia) (highest score of Items 1 to 4); appetite/weight disturbance (highest score of Items 6 to 9); and psychomotor disturbance (highest score of Items 15 and 16). The QIDS-SR16 total score is calculated as the sum of the 9 domain scores. The QIDS-SR16 total score ranges from 0 to 27 with a high score indicating more severe symptoms.
Time Frame: baseline, 12 weeks (LOCF)
Population: only 351 of the 377 subjects had the QIDS-SR16 assessment at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 351
units on a scale | -1.0 (3.23)

3. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the Positive and Negative Syndrome Scale Positive Subscale (PANSS P) Score
Description: The PANSS-P is a subset of items in the PANSS, an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS-P subscale score is the sum of the 7 items and ranges from 7 through 49. A higher score is associated with greater illness severity.
Time Frame: baseline, 12 weeks (LOCF)
Population: only 359 of the 377 subjects had the PANSS-P assessment at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 359
units on a scale | -0.2 (1.16)

4. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the YMRS Total Score -Mania as Assessed by Young Mania Rating Scale (YMRS)
Description: Movement disorders as assessed by Young Mania Rating Scale (YMRS) The YMRS is an 11-item instrument used to assess the severity of mania in subjects with a diagnosis of bipolar disorder. Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score). The YMRS total score is calculated as the sum of the 11 items. The YMRS total score ranges from 0 to 60. Higher scores are associated with greater severity of mania.
Time Frame: Baseline, 12 weeks (LOCF)
Population: only 375 of the 377 subjects had the YMRD assessment at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 375
units on a scale | -1.0 (5.17)

5. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the MADRS Total Score- Depression as Assessed by Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Depression as assessed by Montgomery-Asberg Depression Rating Scale (MADRS) -The MADRS consists of 10 items, each rated on a Likert scale, from 0="Normal" to 6="Most Severe". The MADRS total score is calculated as the sum of the 10 items. The MADRS total score ranges from 0 to 60. Higher scores are associated with greater severity of depression.
Time Frame: baseline ,Week 12 (LOCF)
Population: Only 375 of the 377 subjects had the MADRS assessment at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 375
units on a scale | -1.9 (6.82)

6. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the CGI-BP-S Overall Score- Severity of Illness as Assessed by the Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S)
Description: Severity of illness as assessed by the Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) -The CGI-BP-S overall score is a single value, clinician-rated assessment of overall bipolar illness severity and ranges from 1= 'Normal, not at all ill' to 7= 'Among the most extremely ill patients'. A higher score is associated with greater illness severity.
Time Frame: baseline, week 12 (LOCF)
Population: only 375 of the 377 subjects had the CGI-BP-S overall assessment at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 375
units on a scale | -.31 (1.068)

7. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the CGI-BP-S Mania Score
Description: The CGI-BP-S mania score is a single value, clinician-rated assessment of mania illness severity and ranges from 1=Normal, not at all ill to 7= Among the most extremely ill patients. A higher score is associated with greater illness severity
Time Frame: baseline, week 12 (LOCF)
Population: Only 375 of the 377 subjects had the CGI-BP-S mania assessment at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 375
units on a scale | -0.13 (0.807)

8. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the CGI-BP-S Depression Scale
Description: The CGI-BP-S depression score is a single value, clinician-rated assessment of depression illness severity and range from 1=normal, not at all ill to 7=Among the most extremely ill patients. A higher score is associated with greater illness severity.
Time Frame: baseline, week 12 (LOCF)
Population: only 375 of the 377 subjects had the CGI-BP-S depression assessment at Week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 375
units on a scale | -0.27 (0.969)

9. Secondary Outcome: Change From Baseline to Week 12 (LOCF) in the SDS Total Score
Description: The SDS is a composite of three self-rated items designed to measure the extent to which three major sectors in the patient's life are impaired by depressive symptoms. The SDS total score is calculated as the sum of the 3 items. The SDS total score ranges from 0 to 30. Higher scores are associated with greater severity of global functional impairments. If a subject has not worked/studied at all during the past week for reasons unrelated to the disorder, the SDS total score will be set to missing.
Time Frame: baseline, week 12 (LOCF)
Population: only 297 of the 377 subjects had the SDS total score at week 12 (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 297
units on a scale | -1.4 (5.98)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Lurasidone
Serious Adverse Events (participants affected / at risk) | 14/377
Other Adverse Events (participants affected / at risk) | 51/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=377)
anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (17)
craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
femur fracture (Injury, poisoning and procedural complications) | 1 (1)
intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
depression (Psychiatric disorders) | 4 (4)
mania (Psychiatric disorders) | 2 (2)
bipolar disorder (Psychiatric disorders) | 1 (1)
emotional distress (Psychiatric disorders) | 1 (1)
panic attack (Psychiatric disorders) | 1 (1)
persecutory delusion (Psychiatric disorders) | 1 (1)
accelerated hyertension (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=377)
nausea (Gastrointestinal disorders) | 8 (9)
nasopharyngitis (Infections and infestations) | 13 (14)
headache (Nervous system disorders) | 15 (18)
akathisia (Nervous system disorders) | 12 (13)
insomnia (Psychiatric disorders) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.